CLINICAL TRIAL: NCT02883023
Title: Electrosclerotherapy as a Novel Treatment Option for Capillary Malformations: A Pilot Study
Brief Title: Electrosclerotherapy for Capillary Malformations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sophie Horbach (Other)
Collaborators: IGEA (Industry)
Responsible Party: Sponsor-Investigator, Sophie Horbach, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58824
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Capillary Malformations; Vascular Malformations
Keywords: Bleomycin; Electroporation
MeSH Terms: conditions — Capillary Malformations, Congenital, 1; Vascular Malformations | interventions — Electrochemotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Electrosclerotherapy (Experimental): One region of interest in the capillary malformation (approximately 1.5x1.5cm)will be treated with electrosclerotherapy
  Interventions: Other: Electrosclerotherapy
- Intralesional bleomycin injections (Active Comparator): One region of interest in the capillary malformation will be treated with intralesional bleomycin injections without electroporation
  Interventions: Drug: Intralesional bleomycin injection
- No treatment (No Intervention): One region of interest in the capillary malformation (approximately 1.5x1.5cm)will not be treated.

INTERVENTIONS:
Other: Electrosclerotherapy — Combination of intralesional bleomycin sclerotherapy and electroporation
  Other Names: Electrochemotherapy
  Arms: Electrosclerotherapy
Drug: Intralesional bleomycin injection — Local intralesional injections with bleomycin
  Other Names: bleomycin sclerotherapy
  Arms: Intralesional bleomycin injections

SUMMARY:
Capillary malformations (port-wine stains) consist of abnormally developed capillary blood vessels in the skin. To date, laser therapy is the only widely accepted treatment modality for capillary malformations, but this therapy has a suboptimal effect in approximately 50-60% of patients.

Intralesional bleomycin injections (sclerotherapy) are a common effective treatment option for vascular malformations with blood vessels with larger diameters. However, bleomycin cannot be injected adequately in the small sized vessels of capillary malformations. The use of an electric field over the tissue (electroporation) may solve this problem: it increases cell membrane permeability and therefore promotes localized delivery of drugs, within (endothelial) cells.

Electroporation in combination with bleomycin sclerotherapy ('electrosclerotherapy') may therefore offer new therapeutic options for capillary malformations. This proof of principle study aims to explore the effectiveness, safety and feasibility of this potential treatment option in a within-patient-controlled pilot study.

DETAILED DESCRIPTION:
Capillary malformations are congenital abnormalities of the capillaries in the skin. These abnormally developed blood vessels cause a red color of the skin (also known as 'port-wine stain'),often in combination with a cobble-stone like aspect of the skin. Currently, the only widely accepted treatment option is laser therapy, in which the abnormal blood vessels are targeted with photocoagulation. However, in approximately 50-60% of patients, treatment outcome of laser therapy is suboptimal. Furthermore, re-darkening of the capillary malformation often occurs after laser therapy. Hence, there is a need for an alternative treatment option - especially for treatment-resistant and recurrent capillary malformations.

Intralesional bleomycin injections (sclerotherapy) are a common treatment option for vascular malformations of blood vessels and lymphatic vessels with a larger diameter (venous and lymphatic malformations). According to the literature, this treatment is effective in approximately 80-90% of patients. Unfortunately, the diameter of capillary blood vessels is too small, and therefore adequate localized injections of bleomycin are not possible in capillary malformations.

'Electroporation' is a physical phenomenon that causes an alteration of the structure of cell membranes through the exposure of cells to a short but intense electric field; this modification of the cell membrane increases its permeability. After electroporation, molecules that normally do not cross the cell membrane, either by diffusion or by active transport, can reach the intracellular environment. Therefore, electroporation is an ideal method for localized drug delivery, in particular for localized bleomycin delivery.

The combination of electroporation and bleomycin is already used in a variety of skin lesions, such as squamous cell carcinoma, with a surprisingly high rate of complete remission. Especially in vascular tumors, such as Kaposi sarcoma, there is an extremely high percentage of complete remission (90%), since the combination of bleomycin and electroporation causes a 'vascular lock' and intravascular thrombosis of tumor vascularization, leading to tumor regression.

This phenomenon (intravascular thrombosis and lesion regression) is exactly the intended effect of capillary malformation treatment.

The investigators therefore hypothesize that intralesional bleomycin injections combined with electroporation (electrosclerotherapy) can be an alternative treatment option for capillary malformations. This proof of principle study aims to explore the feasibility of this potential treatment option in a small patient sample.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥1 completely or partially hypertrophic capillary malformation not exclusively located in the skin of the face, the skin overlying joints or in mucosal tissue
* Age ≥ 18 years
* Fitzpatrick skin type 1-3 without evident sun tan

Exclusion Criteria:

* Pregnant or breastfeeding women
* Women with childbearing potential not using contraception
* Patients with chronic renal dysfunction of GFR <50 ml/minute
* Patients with chronic pulmonary dysfunction, active pulmonary infections or previous bleomycin lung toxicity
* Patients with ataxia teleangiectasia
* Patients with previous allergic reactions to bleomycin
* Patients who already received the maximum dose of bleomycin (400 mg or 400000 IU/m2)
* Patients with implanted electrical devices such as pacemakers or ICD's
* Patients with clinically manifested arrhythmia
* Patients with epilepsy
* Patients who are not able to return to the hospital for follow-up visits
* Patients who are likely not able to understand the terms and risks of the study (e.g. cognitive impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer global assessment of capillary malformation (POSAS instrument) | 7 weeks
  Change in patient and observer assessment of vascularity, pigmentation, thickness, pliability, relief, surface area and general opinion.

SECONDARY OUTCOMES:
Adverse events | 7 weeks
  Any adverse event or serious adverse event occurring after intervention
Colorimetry | 7 weeks
  Change in color of capillary malformation in relation the contralateral healthy skin
Optical imaging (laser speckle imaging) | 7 weeks
  Change in blood perfusion measured with non invasive imaging using light

CONTACTS AND LOCATIONS:
Overall Officials: Chantal M van der Horst, MD PhD, Principal Investigator — Academic Medical Center (AMC)
Locations (1):
- Academic Medical Center (AMC), Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horbach SER, Wolkerstorfer A, Jolink F, Bloemen PR, van der Horst CMAM. Electrosclerotherapy as a Novel Treatment Option for Hypertrophic Capillary Malformations: A Randomized Controlled Pilot Trial. Dermatol Surg. 2020 Apr;46(4):491-498. doi: 10.1097/DSS.0000000000002191. PMID 31574025
- [Derived] Horbach SER, Wolkerstorfer A, de Bruin DM, Jansen SM, van der Horst CMAM. Electrosclerotherapy for capillary malformations: study protocol for a randomised within-patient controlled pilot trial. BMJ Open. 2017 Nov 14;7(11):e016401. doi: 10.1136/bmjopen-2017-016401. PMID 29138199